CLINICAL TRIAL: NCT03090269
Title: Pilot Study to Evaluate the Benefits and the Risks of Methylphenidate for the Treatment of Cocaine Dependence
Brief Title: Methylphenidate for Cocaine Dependence
Acronym: ANRS STIMAGO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: feasibility reasons.
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Hopital Paul Brousse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS STIMAGO; 2013-002996-16 (EudraCT Number)
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Substance-Related Disorders
Keywords: cocaine; methylphenidate; psychostimulant; ADHD; effective dose; pharmacokinetics; crack
MeSH Terms: conditions — Substance-Related Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: open-label, single site, national, pilot study, non-comparative before/after
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylphenidate pill (Experimental): 18 mg tablets with a 3-week titration phase to a maximum dose of 108 mg per day, orally
  Associated with phone interviews every month, urine drug toxicologies and blood sampling (PK/PD)
  Interventions: Drug: Methylphenidate Pill

INTERVENTIONS:
Drug: Methylphenidate Pill — 3-month follow-up to study the effective dose as a treatment for cocaine dependence in toxicity and reduction in cocaine use
  Other Names: Concerta

SUMMARY:
This phase II pilot study aims at evaluating the benefits and the risks of methylphenidate (Concerta®) for the treatment of cocaine/crack dependence in terms of cocaine/crack use reduction and adverse events.

DETAILED DESCRIPTION:
Patients will receive pharmacotherapy based on methylphenidate (18 mg per tablet) with a 3-week titration phase to a maximum dose of 108 mg per day, with a weekly follow-up during 3 months. Socio-demographic and behavioral data will be collected through phone interviews every month. During medical visits, self-administered and clinical questionnaires will collect clinical and behavioral data. Urine drug toxicologies and blood sampling will be performed to gather biological, pharmacokinetic and pharmacodynamic data.

This study should identify an effective response-dose of methylphenidate for people with a cocaine use disorder. The methylphenidate should be effective to reduce cocaine use in cocaine-dependent individuals with a good tolerability. The results of pharmacokinetic and pharmacodynamic analyses will give us the effective dose of methylphenidate and some information on toxicity to adapt the surveillance in a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cocaine/crack/amphetamine derivate dependence using Diagnostic and Statistical Manual of Mental Disorders (DSM V) (and International Classification of Diseases (ICD 10)) and willing to be abstinent.
* Having a cocaine/crack positive urinary test.
* Effective contraception for women of childbearing age.
* Willing to participate.
* Registered at social insurance/security.
* Being able to give consent.
* Reachable by telephone.

Exclusion Criteria:

* Dependence on alcohol and/or other substances.
* Hypersensitivity to the active compound methylphenidate or to filler.
* Glaucoma.
* Phaeochromocytoma
* Family history or diagnosis of Gilles de la Tourette syndrome.
* During treatment with non-selective, irreversible monoamine oxidase (MAO) inhibitors.
* History of hyperthyroidism or of thyrotoxicosis.
* Preexisting cardiovascular problems including severe hypertension, heart failure, arterial occlusive disease, angina, haemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening arrythmias and channelopathies, (disorders caused by the dysfunction of ionic channels).
* Preexisting cerebrovascular disorders, cerebral aneurism, vascular abnormalities including vasculitis or stroke.
* Diagnosis or history of severe depression, anorexia nervosa/anorexic disorders, suicidal tendencies, psychotic symptoms, severe mood disorders, mania, schizophrenia, psychopathic/borderline personality disorder
* Diagnosis or history of severe and episodic (Type I) Bipolar (affective) Disorder (that is not well-controlled)
* Suicidal tendencies or characterized suicidal syndrome.
* Pregnancy, breast-feeding or absence of any contraception for female participants.
* Unstabilized psychiatric comorbidity likely to compromise adherence to treatment.
* Comorbidity or handicap likely to corrupt evaluation.
* Organic pathology severe enough according to the investigator, likely to comprise adequate surveillance during the trial.
* Patient about to leave the area for a period of time preventing his/her adequate participation in the trial.
* Insufficient motivation.
* Participation in another clinical trial with an on-going exclusion period at the time of the pre-inclusion visit.
* Lack of medical insurance.
* Unreachable by phone.
* Patient on mandatory treatment.
* Patient with legal incapacity (under guardianship or curatorship)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Cocaine use | Evaluated through the study: during the titration phase (day 1, day 4, day 8, day 11, day 15, day 18) and then at the week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11 and week 12
  Difference between weekly cocaine use at M0 and M3 based on the patient self-reports and urinalysis

SECONDARY OUTCOMES:
Side effects using the Drug Effects questionnaire (DEQ) | Evaluated at the week 1, week 2, week 4, week 9 and week 12
  Number of perceived side effects of methylphenidate with the Drug Effects questionnaire (DEQ)
Craving using the Cocaine Craving Questionnaire (CCQ 10-item) | Evaluated during the titration phase (day 1, day 4, day 8, day 11, day 15, day 18) and then at each visit of the two last months (1 visit a week for 2 months)
  Cocaine craving with the Cocaine Craving Questionnaire (CCQ 10-item)
Abstinence (urinalysis) | Evaluated during the titration phase (day 1, day 8, day 15, day 18) and then at the week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11 and week 12
  Cocaine abstinence with urinalysis
Risk practices using the Blood Borne Virus Transmission Risk Assessment Questionnaire (BBV-TRAQ) | Evaluated at the week 1, week 4, week 9 and week 12
  Reduction in Hepatitis C (HCV) risk practices, unsafe sex, sharing syringes - Blood Borne Virus Transmission Risk Assessment Questionnaire (BBV-TRAQ)
Psychiatric symptoms - Depression using the Center for Epidemiologic Studies - Depression Scale (CES-D) | Evaluated at the week 1, week 4, week 9 and week 12
  Reduction in psychiatric symptoms with the Center for Epidemiologic Studies - Depression Scale (CES-D)
Psychiatric symptoms - Attention/Deficit using the attention-deficit/hyperactivity disorder Scale (ADHD) | Evaluated at the week 1, week 4, week 9 and week 12
  Reduction in psychiatric symptoms with the attention-deficit/hyperactivity disorder Scale (ADHD)
Psychiatric symptoms - Sensation Seeking using the 6-item Sensation Seeking Scale (SSQ 6-item) | Evaluated at the week 1, week 4, week 9 and week 12
  Reduction in psychiatric symptoms with the 6-item Sensation Seeking Scale (SSQ 6-item)
Criminal behaviors | Evaluated at the week 1, week 4, week 9 and week 12
  Reduction in self-reported criminal behaviors by questionnaire
Quality of life using the the 12-Item Short Form Health Survey (SF-12) | Evaluated at the week 1, week 4, week 9 and week 12
  Increase of quality of life score with the 12-Item Short Form Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Amine Benyamina, Pr, Principal Investigator — Hôpital Paul Brousse APHP - France
Locations (1):
- Hôpital Paul Brousse, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor of the study — http://anrs.fr